CLINICAL TRIAL: NCT05076435
Title: Restrictive Fluid Administration vs. Standard of Care in Emergency Department Sepsis Patients - a Multicenter, Randomized Clinical Feasibility Trial (REFACED Sepsis)
Brief Title: Restrictive Fluid Administration vs. Standard of Care in Emergency Department Sepsis Patients
Acronym: REFACED Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marie Kristine Jessen, MD (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other); Viborg Regional Hospital (Other); Randers Regional Hospital (Other)
Responsible Party: Sponsor-Investigator, Marie Kristine Jessen, MD, Principal Investigator, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECEM0001; 2021-000224-35 (EudraCT Number); 1-10-72-163-21 (Other: The Committee on Health Research Ethics, Central Denmark Region)
Record Dates: First submitted 2021-09-11; First posted 2021-10-13 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Sepsis
Keywords: Sepsis; Hypotension; IV fluid therapy; Fluid resuscitation; Emergency Department; Crystalloids
MeSH Terms: conditions — Sepsis; Hypotension; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive fluid administration (Experimental): No IV fluids unless one of the extenuating circumstances occur;
  1. In case of severe hypoperfusion or severe circulatory impairment defined by either: 1) Lactate≥4 mmol/L, 2) Hypotension (systolic BP < 90 mmHg), 3) Mottling beyond the kneecap (mottling score >2) OR 4) Urinary output<0.1 mL/kg bodyweight/h (only in the first 4hrs after randomization) then a bolus of 250 ml of IV crystalloid solution may be given followed by re-evaluation
  2. In case of overt fluid losses (e.g. vomiting, large aspirates,) IV fluid may be given to correct for the loss, but not above the volume lost.
  3. In case the oral/enteral route for water or electrolyte solutions is contraindicated or has failed, IV fluids may be given to:
     Correct dehydration or electrolyte deficiencies Ensure a total fluid input of 1 L in 24hrs
  4. IV fluids may be given as carrier for medication, but with lowest possible volume
  Interventions: Drug: Isotonic crystalloids
- Usual care (standard care) (Active Comparator): There will be no upper limit for the use of either IV or oral/enteral fluids
  1. IV fluids should be given in the case of hypoperfusion or circulatory impairment and should be continued as long as hemodynamic variables improve including static or dynamic variable(s) as chosen by the clinicians. These criteria are based on the Surviving Sepsis Campaign guideline.
  2. IV fluids should be given as maintenance if the ICU has a protocol recommending maintenance fluid
  3. IV fluids should be given to substitute expected or observed loss, dehydration or electrolyte derangements
  Interventions: Drug: Isotonic crystalloids

INTERVENTIONS:
Drug: Isotonic crystalloids — Types of fluids in both intervention groups:
  * Fluids used for electrolyte disturbances: Fluids should be chosen to substitute the specific deficiency
  * Fluids given to substitute overt loss: Isotonic crystalloids are to be used. If large amounts of ascites are tapped, then human albumin may be used.
  * Blood products are only to be used on specific indications including severe bleeding, severe anaemia and prophylactic in case of severe coagulopathy.

SUMMARY:
This is an investigator-initiated, multicenter, randomized, parallel-group, open-labeled, feasibility trial investigating volumes of fluid within 24 hours in 124 patients with sepsis allocated to two different IV fluid regimens enrolled at three emergency departments in Central Region Denmark. The primary outcome is total intravenous, crystalloid fluid volume within 24 hours and key secondary outcomes include protocol violations, total fluids (intravenous and oral) within 24 hours, SAEs/SUSARs, and inhospital-, 30- and 90-day mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Sepsis is common in emergency department (ED) patients. Traditionally, intravenous (IV) fluids are used to optimise the circulation, and the use of higher volumes is recommended by international guidelines, but there are no recommendations for sepsis without hypotension or shock. Studies in septic shock seem to favour fluid restriction. Whether this is true in sepsis without hypotension/shock is unknown.

OBJECTIVES:

The aim of the REFACED Sepsis trial is to test if an IV fluid restrictive protocol in ED patients with sepsis is feasible, i.e., if the protocol decreases the IV fluid volumes administered.

DESIGN:

REFACED Sepsis is a multicenter, randomized, parallel-group, open-labeled, feasibility trial

POPULATION:

ED patients with sepsis expected to be admitted for ≥ 24 hours

EXPERIMENTAL INTERVENTION:

In the IV fluid restriction group no IV fluids should be given unless one of the below mentioned occurs;

A fluid bolus of 250 ml isotonic crystalloid may be given within 15 minutes if one of the following occurs (hypoperfusion criteria):

* Lactate concentration ≥ 4 mmol/l (arterial or venous blood gas/blood sample)
* Hypotension (systolic BP < 90 mmHg)
* Mottling beyond edge of kneecap (i.e., Mottling score >2)53
* Severe oliguria, i.e., diuresis < 0.1 ml/kg/h, during the first 4 hours of admission

All patients will be ensured min. 1 L of oral/intravenous fluids in 24 hours and electrolytes can be corrected.

CONTROL INTERVENTION:

In the usual care group there will be no upper limit for the use of IV fluids.

OUTCOMES:

The primary outcome is 24-hour intravenous crystalloid fluid administration. Key secondary outcomes are: Feasibility measures: Number of patients with major protocol violations, Number of patients screened vs included, Time from admission to inclusion, Number of patients lost to follow up in terms of 24-hour fluids, Accumulated serious adverse reactions and events (SAEs + Suspected Unexpected Serious Adverse Reaction (SUSARs)) within 48 hours in-hospital, Total fluids (oral and intravenous) at 24 hours,

TRIAL-SIZE:

124 patients will be randomized to restrictive fluid administration or usual care within 24 hours of randomization

ELIGIBILITY:
Inclusion Criteria: All of the below must be fulfilled:

1. Unplanned emergency department admission
2. Age ≥ 18 years
3. Sepsis defined as

   1. suspected infection by the treating clinician AND
   2. blood cultures drawn AND
   3. IV antibiotics administered or planned AND
   4. An infection related increase of SOFA*-score ≥ 2 from baseline
4. Expected hospital stay > 24 hours as deemed by treating clinician

   * Sequential Organ Failure Assessment (SOFA) Score

Further more the patient must fulfill criteria for enrollment in an acute study according to Danish law

Exclusion Criteria: We will exclude patients fulfilling any of following exclusion criteria:

1. ≥ 500 ml of fluids given prior to randomization
2. Invasively ventilated or vasopressors initiated at the time of screening
3. Known or suspected severe bleeding judged by the treating clinician
4. Known or suspected pregnancy (women aged <45 years will have a pregnancy test performed before enrollment)
5. Prior enrollment in the trial
6. Patients, who the clinician expect not to survive the next 24-hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-03-19 (Actual)

PRIMARY OUTCOMES:
24-hour crystalloid iv. fluids | 24 hours from randomization
  total amount of all administered intravenous, crystalloid fluids within 24 hours of randomization

SECONDARY OUTCOMES:
Protocol violations | 24 hours from randomization
  Feasibility measure: Number of patients with major protocol violations
Screened-vs.-randomized-ratio | Through study completion, an average of 1 year
  Feasibility measure: Number of patients screened vs included
Time to inclusion | Through study completion, an average of 1 year
  Feasibility measure: Time from admission to inclusion/randomization (hours)
Lost-to-follow-up-rate | 24 hours from randomization
  Feasibility measure: Number of patients lost to follow up in terms of 24-hour fluids
Accumulated serious adverse reactions (SARs + SUSARs) | 7 days from randomization
  Feasibility measure: Accumulated serious adverse reactions and events (SAEs + SARs+ SUSARs) within 7 days in-hospital
Total 24-hour fluids | 24 hours from randomization
  Total fluids (oral and intravenous) at 24 hours
Mortality | Total of 90-days
  In-hospital, 30- and 90-days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marie K Jessen, MD, Principal Investigator — Research Center for Emergency Medicine, Department of Clinical Medicine, Aarhus University and Aarhus University Hospital, Denmark
Locations (3):
- Denmark (3):
  - Department of Emergency Medicine, Aarhus University Hospital, Aarhus, Central Jutland
  - Department of Emergency Medicine, Regional Hospital Randers, Randers, Central Jutland
  - Department of Emergency Medicine, Regional Hospital Viborg, Viborg, Central Jutland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jessen MK, Andersen LW, Thomsen MH, Kristensen P, Hayeri W, Hassel RE, Messerschmidt TG, Solling CG, Perner A, Petersen JAK, Kirkegaard H. Restrictive fluids versus standard care in adults with sepsis in the emergency department (REFACED): A multicenter, randomized feasibility trial. Acad Emerg Med. 2022 Oct;29(10):1172-1184. doi: 10.1111/acem.14546. Epub 2022 Aug 5. PMID 35652491
- [Derived] Jessen MK, Andersen LW, Thomsen MH, Kristensen P, Hayeri W, Hassel RE, Perner A, Petersen JAK, Kirkegaard H. Restrictive Fluid Administration vs. Standard of Care in Emergency Department Sepsis Patients (REFACED Sepsis)-protocol for a multicenter, randomized, clinical, proof-of-concept trial. Pilot Feasibility Stud. 2022 Mar 29;8(1):75. doi: 10.1186/s40814-022-01034-y. PMID 35351214